CLINICAL TRIAL: NCT07241858
Title: Clinicolaboratory Predictors of Outcome in Children With Encephalitis
Acronym: encephalitis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Mostafa Sayed Mostafa, Assistant Lecturer, Assiut University
Other Study IDs: pediatric encephalitis
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Encephalitis in Children; Encephalitis
MeSH Terms: conditions — Encephalitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with encephalitis
  Interventions: Diagnostic Test: CSF analysis and culture including S100B,Neuron Specific Enolase(NSE)

INTERVENTIONS:
Diagnostic Test: CSF analysis and culture including S100B,Neuron Specific Enolase(NSE) — CSF analysis and culture including S100B,Neuron Specific Enolase(NSE)

SUMMARY:
. A glycolytic enzyme called enolase is primarily found in neurons. A dimeric isoform of enolase called neuron-specific enolase (NSE) exists. It can be found in neurons, platelets, erythrocytes, and other neuroectodermal cells.It is one of the laboratory biomarkers that could be investigated in cases of encephalopathy, which can be found in both blood and cerebrospinal fluid, might be a helpful biomarker for determining brain injury prognosis and neuronal damage.(4) High S-100beta levels were associated with higher intensive care unit mortality and represented the strongest independent predictor of intensive care unit survival, whereas neuron-specific enolase (NSE) and the Glasgow Coma Scale failed to predict fatal outcome.(5) (NSE) and S100B are important as a diagnostic and a prognostic value in pediatric encephalopathy which is common and is potentially life threatening, previous studies were done worldwide to detect its diagnostic and prognostic value in acute encephalopathy among adult and pediatric age groups.(4) ,so we asses (NSE) and S100B to detect the the out come of acute encephalopathy

DETAILED DESCRIPTION:
Acute encephalopathy is the generic term for acute brain dysfunction caused by various agents, such as infection, metabolic disease, hepatic or renal dysfunctions, and hypertension;causing change in mental status that affects cognition or level of alertness in the patient. The pathological substrate of acute encephalopathy is diffuse or widespread non-inflammatory brain edema..(1) The key for establishing evidence of central nervous system (CNS) inflammation is the analysis of CSF. Lumbar puncture (LP) is often excessively delayed, primarily due to performing brain imaging to exclude raised intracranial pressure. Not all patients need imaging before LP, and consensus guidelines suggest a few clear indications for imaging. If these are present, then either a computed tomography (CT) scan or, ideally, magnetic resonance imaging (MRI) should be obtained urgently. Following this, if there are no radiological contraindications, LP should be performed as soon as possible. Brain imaging serves three purposes: to look for changes of encephalitis, to exclude alternative diagnoses, and to assess patency of the basal cisterns and an absence of mass effect so that LP can proceed.(2) Biochemical markers can be used in addition to neuroimaging techniques to evaluate the extent of brain injuries and to enable earlier diagnosis and faster intervention. Among the potential biomarkers of brain injuries, neuron-specific enolase (NSE) and S100B are the most frequently studied and were shown to be the most promising.(3).

ELIGIBILITY:
Inclusion Criteria:

* 1. Pediatric population aged 1month to 18 years.

  * Decreased level of consciousness, personality change, or psychiatric manifestations lasting >24 h (in toddlers and infants, may present as increased irritability or lethargy)
  * No alternative diagnosis to explain presentation
  * Seizure (new onset)
  * Fever (≥38.0°C)
  * Focal neurologic findings (new onset)
  * CSF WBC ≥5/mm3

Exclusion Criteria:

* 1. Neonates and adults ( <1 month or >18 years) 2. If they had a diagnosis of delirium or encephalopathy secondary to sepsis, toxins,renal ,hepatic or metabolic causes (hypoglycemia, electrolyte disturbances

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Pediatric population aged 1month to 18 years.
  * Decreased level of consciousness, personality change, or psychiatric manifestations lasting >24 h (in toddlers and infants, may present as increased irritability or lethargy)
  * No alternative diagnosis to explain presentation
  * Seizure (new onset)
  * Fever (≥38.0°C)
  * Focal neurologic findings (new onset)
  * CSF WBC ≥5/mm3
  * Acute abnormality on brain MRI
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
To asses clinical ,radiological laboratory biomarkers ( CSF Neuron-Specific Enolase and S100B )as outcome predictors of encephalitis | 1 month
  To asses clinical ,radiological laboratory biomarkers ( CSF Neuron-Specific Enolase and S100B )as outcome predictors of encephalitis

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Makovec M, Skitek M, Simnovec L, Jerin A. Neuron-Specific Enolase and S100B as Biomarkers of Ischemic Brain Injury During Surgery. Clin Pract. 2025 Apr 3;15(4):74. doi: 10.3390/clinpract15040074. PMID 40310303
- [Background] Aneja S, Sharma S. Diagnosis and Management of Acute Encephalitis in Children. Indian J Pediatr. 2019 Jan;86(1):70-75. doi: 10.1007/s12098-018-2775-0. Epub 2018 Sep 19. PMID 30232787
- [Background] Shiihara T, Miyake T, Izumi S, Watanabe M, Kamayachi K, Kodama K, Nabetani M, Ikemiyagi M, Yamaguchi Y, Sawaura N. Serum and cerebrospinal fluid S100B, neuron-specific enolase, and total tau protein in acute encephalopathy with biphasic seizures and late reduced diffusion: a diagnostic validity. Pediatr Int. 2012 Feb;54(1):52-5. doi: 10.1111/j.1442-200X.2011.03454.x. Epub 2011 Oct 30. PMID 21883688